CLINICAL TRIAL: NCT02848443
Title: Phase I Dose-escalation of S 95005 (TAS-102) in Combination With Oxaliplatin in Metastatic Colorectal Cancer
Brief Title: Study of S 95005 in Combination With Oxaliplatin in Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-95005-001; 2015-004894-34 (EudraCT Number)
Record Dates: First submitted 2016-02-24; First posted 2016-07-28 (Estimated); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; oxaliplatin; dose-escalation; Lonsurf; nivolumab; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Trifluridine; Oxaliplatin; Bevacizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S 95005 + oxaliplatin (+/- bevacizumab or nivolumab) (Experimental)
  Interventions: Drug: Trifluridine/tipiracil hydrochloride (S 95005); Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil hydrochloride (S 95005) — Film-coated tablets containing 15mg of trifluridine and 7.065mg of tipiracil hydrochloride, or 20mg of trifluridine and 9.42mg of tipiracil hydrochloride, given orally at the dose of 25 or 30 or 35 mg/m2/dose, until unacceptable toxicity according to the investigator, disease progression or patient withdrawal.
Drug: Oxaliplatin — Concentrate for solution for infusion containing 5mg/ml of oxaliplatin, administered intravenously at the dose of 65 to 85 mg/m2, until unacceptable toxicity according to the investigator, disease progression or patient withdrawal.
Drug: Bevacizumab — Concentrate for solution for infusion containing 25mg/ml of bevacizumab, administered intravenously at the dose of 5 mg/kg, until unacceptable toxicity according to the investigator, disease progression or patient withdrawal.
Drug: Nivolumab — Concentrate for solution for infusion containing 10mg/ml of nivolumab, administered intravenously at the dose of 3 mg/kg, until unacceptable toxicity according to the investigator, disease progression or patient withdrawal.

SUMMARY:
The main purpose of this study is to assess the safety and tolerability and to determine the recommended phase 2 dose of S 95005 given in combination with oxaliplatin in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a one-arm study, which will be conducted in 2 parts:

* A dose-escalation part to determine the Maximum Tolerated Dose (MTD) of S 95005 in combination with oxaliplatin.
* An expansion part in patients treated at the recommended dose defined in the dose escalation part of this study to evaluate the safety, PK, and preliminary efficacy of S 95005 in combination with oxaliplatin and either bevacizumab or nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Histologically confirmed metastatic colorectal cancer pretreated by at least one line of standard chemotherapy.
* Restaging scan within 28 days before the first study drug intake.
* During the dose-escalation part, patient must have at least one evaluable or measurable metastatic lesion; and during the expansion part, patient must have at least one measurable metastatic lesion.
* Life expectancy of more than 3 months.
* Performance status Eastern Cooperative Oncology Group (ECOG): 0-1.
* Adequate bone marrow, liver, and kidney function.
* For patients who will receive bevacizumab: coagulation parameters in normal limit or in therapeutic limit for patients treated with anticoagulant.
* For patients who will receive nivolumab: patients eligible for tumour biopsy and who agree to have two sequential biopsies during the study.
* Women of childbearing potential must have a negative pregnancy test. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use highly effective birth control method. Women and female partners using hormonal contraceptive must also use a barrier method.
* Capacity to take oral tablet(s) without difficulty.
* Has provided written informed consent.
* Is willing and able to comply with scheduled visits and study procedures.

Exclusion Criteria:

* Grade 2 or higher peripheral neuropathy.
* During expansion part, patients who had recurrence during or within 6 months of completion of the adjuvant chemotherapy with oxaliplatin.
* Patients with brain metastases or leptomeningeal metastasis.
* Other malignancy within the last 3 years (except for basal cell carcinoma or a non-invasive/in situ cervical cancer)
* Has had certain other recent treatment e.g. major surgery, field radiation, participation in another interventional study, within the specified time frames prior to study drug administration.
* Certain serious illnesses or serious medical conditions
* For patients who will receive bevacizumab: history of allergic reactions/hypersensitivity to bevacizumab, to any components used in the formulation, to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies.
* Grade 3 or higher hypersensitivity reaction to oxaliplatin or garde 1-2 hypersensitivity reaction to oxaliplatin not controlled with premedication.
* Patient previously treated by S 95005 or history of allergic reactions attributed to compounds of similar composition to S 95005 or any of its excipient. Patient with hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Any condition that, in the judgment of the Investigator, may affect the patient's ability to understand and sign the informed consent and fully comply with all study procedure.
* Pregnancy or breast feeding.
* For patients planned to receive nivolumab:

  * Patients with active autoimmune disease or history of clinically severe autoimmune disease.
  * Patients with a condition requiring systemic treatment with either corticosteroids (> 20 mg daily prednisone equivalent) or other immunosuppressive medications within the specified time frames prior to first study drug intake.
  * Prior treatment with anti-PD-1, anti-PD-L1, anti-programmed cell death ligand-2, anti-CD137, anti-OX-40, anti-CD40, anti-cytotoxic T lymphocyte-associated antigen-4 antibodies (CTLA-4), or any other immune checkpoint inhibitors.
  * Prior events of immune-mediated pneumonitis, immune-mediated colitis, immune-mediated hepatitis, immune-mediated endocrinopathies, immune-mediated nephritis and renal dysfunction, immune-mediated rash, immune-mediated encephalitis.
  * Allergic reactions/hypersensitivity to nivolumab or any components used in its formulation or previous severe hypersensitivity reaction to treatment with another monoclonal antibody.
  * Has a known history of active tuberculosis (Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of S95005 when given in combination with oxaliplatin | up to 4 weeks after the first treatment administration
Dose Limiting Toxicity (DLT) of S95005 when given in combination with oxaliplatin | up to 4 weeks after the first treatment administration
Number of participants with adverse events as a measure of safety and tolerability for S95005-oxaliplatin. | through study completion, an average of 9 months
  Adverse event reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03
Changes in standard hematology as a measure of safety and tolerability for S95005-oxaliplatin | through study completion, an average of 9 months
Changes in biochemistry as a measure of safety and tolerability for S95005-oxaliplatin | through study completion, an average of 9 months
Changes in coagulation as a measure of safety and tolerability for S95005-oxaliplatin | through study completion, an average of 9 months
Changes in urinalysis as a measure of safety and tolerability for S95005-oxaliplatin | through study completion, an average of 9 months
Changes in vital signs as a measure of safety for S95005-oxaliplatin | through study completion, an average of 9 months
  Vital sign measurements will include temperature, systolic and diastolic blood pressure, heart rate, and respiratory rate.
Changes in ECOG (Eastern Cooperative Oncology Group) performance status as a measure of safety and tolerability for S95005-oxaliplatin | through study completion, an average of 9 months

SECONDARY OUTCOMES:
Antitumor activity assessed by RECIST (Response Evaluation Criteria in Solid Tumors) and CEA (Carcinoembryonic Antigen) | through study completion, an average of 9 months
Number of participants with adverse events as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
  Adverse event reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03
Changes in standard hematology as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
Changes in biochemistry as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
Changes in coagulation as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab. | through study completion, an average of 9 months
Changes in urinalysis as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
Changes in vital signs as a measure of safety for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
  Vital sign measurements will include temperature, systolic and diastolic blood pressure, heart rate, and respiratory rate.
Changes in ECOG (Eastern Cooperative Oncology Group) performance status as a measure of safety and tolerability for S95005-oxaliplatin + bevacizumab or nivolumab. | through study completion, an average of 9 months
PDL-1 expression, tumour-infiltrating CD8 T cell density, for S95005-oxaliplatin + nivolumab | up to 8 weeks after the first treatment administration
  Tumour biopsy at baseline and at the end of Cycle 4

OTHER OUTCOMES:
Circulating protein biomarkers analysis | through study completion, an average of 9 months
  Samples collected at C1D1 (day 1 of cycle 1) and at withdrawal will be subjected to proteomic analysis for identification of potential predictive and resistance biomarkers for S 95005 and/or oxaliplatin response or biological activity.
Circulating tumour DNA analysis | day 1 of cycle 1 (each cycle is 28 days)
  Samples collected at C1D1 will be subjected to genomic analysis to study mutations currently observed in colorectal cancer
Circulating protein biomarkers in relation to ICD (immune cell death) | through study completion, an average of 9 months
  Samples collected at C1D1, C2D1, C3D1 and C5D1 pre-dose then every 4 cycles will be subjected to proteomic analysis to measure immune cell death (ICD) biomarkers potentially induced by the treatment S95005-oxaliplatin + nivolumab.
Peripheral blood mononuclear cells | up to 10 weeks after the first treatment administration
  Samples collected at C1D1 and C5D1 will be subject to analysis for identification of lymphocytes cells phenotypes, for S95005-oxaliplatin + nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: Josef Tabernero, Prof, Principal Investigator — Vall d'Hebron University Hospital, Institute of Oncology (VHIO)
Locations (24):
- Allgemeines Krankenhaus - Universitätskliniken Klinische Abteilung für Onkologie, Vienna, Austria
- France (5):
  - CHU de la Timone Hépato-Gastro-Entérologie - Oncology Digestive, Marseille
  - Hôpital Saint-Antoine Service d'Oncologie Médicale, Paris
  - La Pitié Salpêtrière Centre Investigation clinique Paris Est, Paris
  - Centre Eugène Marquis Service d'Oncologie Médicale, Rennes
  - Institut Gustave Roussy DITEP, Villejuif
- Germany (5):
  - St. Josef-Hospital, Klinikum der Ruhr-Universität Bochum Abteilung für Hämatologie und Onkologie, Bochum
  - Universitätsklinikum Hamburg-Eppendorf II. Medizin. Klinik und Poliklinik (Onkologie, Hämatologie), Hamburg
  - Klinikum der Universität München Campus Großhadern, Medizinische Klinik und Poliklinik III, München
  - Universitätsklinikum Ulm Zentrum für Innere Medizin, Klinik für Innere Medizin I, Ulm
  - Klinikum Wolfsburg Medizinische Klinik II, Wolfsburg
- Hungary (3):
  - Magyar Honvedseg Egeszsegugyi Kozpont Onkologiai Osztaly, Budapest
  - Semmelweis Egyetem I. sz. Belgyogyaszati Klinika - Klin. Farmakologiai Reszleg, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati-Onkologiai O. Es Klin. Farmakologiai O., Budapest
- Italy (3):
  - ARNAS - Azienda Ospedaliera Garibaldi - Nesima Struttura Complessa di Oncologia Medica, Catania
  - Ist.Scientifico Romagnolo per lo Studio e la Cura dei Tumori Department of Clinical Oncology, Meldola
  - Policlinico G.B. Rossi A.O.U.I. di Verona U.O.C. di Oncologia, Verona
- Spain (6):
  - ICO Badalona. H. Germans Trials y Pujol - Servicio de Oncología médica, Badalona
  - H. Valle de Hebrón - Servicio de Oncología - (VHIR), Barcelona
  - Hospital Unviersitario Gregorio Marañon - Servicio de Oncología Médica, Madrid
  - H. Univ. Ramon y Cajal - Servicio de Oncología Medica, Madrid
  - H. Uni. Madrid Sanchinarro - CIOCC Servicio de Oncología, Madrid
  - H. Clinico de Valencia INCLIVA - Departamento de Hematologia y Oncologia Medica 8ª planta, Valencia
- Christie Hospital NHS Foundation Trust GI & Endocrine, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Bordonaro R, Calvo A, Auriemma A, Hollebecque A, Rubovszky G, Saunders MP, Papai Z, Prager G, Stein A, Andre T, Argiles G, Cubillo A, Dahan L, Edeline J, Leger C, Cattan V, Fougeray R, Amellal N, Tabernero J. Trifluridine/tipiracil in combination with oxaliplatin and either bevacizumab or nivolumab in metastatic colorectal cancer: a dose-expansion, phase I study. ESMO Open. 2021 Oct;6(5):100270. doi: 10.1016/j.esmoop.2021.100270. Epub 2021 Sep 20. PMID 34547581
- [Derived] Argiles G, Andre T, Hollebecque A, Calvo A, Dahan L, Cervantes A, Leger C, Amellal N, Fougeray R, Tabernero J. Phase I dose-escalation of trifluridine/tipiracil in combination with oxaliplatin in patients with metastatic colorectal cancer. Eur J Cancer. 2019 May;112:12-19. doi: 10.1016/j.ejca.2019.01.101. Epub 2019 Mar 16. PMID 30889492
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/